CLINICAL TRIAL: NCT06013345
Title: Conventional Vs. Optimised Periprocedural Analgosedation Vs. Total Intravenous Anaesthesia for Pulsed-field Ablation: a Randomised Controlled Trial
Brief Title: COnventional Vs. Optimised PERiprocedural Analgosedation Vs. Total IntraVEnous Anaesthesia for Pulsed-Field Ablation (COOPERATIVE-PFA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Marek Hozman, MD, PhD, Principal investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Coopertaive-PFA
Record Dates: First submitted 2023-08-17; First posted 2023-08-28 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: Analgosedation; Remimazolam; Atrial Fibrillation; Pulsed field ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — remimazolam; Propofol

STUDY DESIGN:
Intervention Model Description: Study arms, analgosedation and TIVA protocols:
  1. Conventional propofol analgosedation (arm P): current standard practice in most centres, a combination of short-acting benzodiazepine (midazolam) at the beginning, short-acting opioid (sufentanil in this study) and propofol boluses before and during the application of ablation pulses with unsecured airway
  2. Optimised continuous intravenous analgosedation (arm R): ultrashort-acting benzodiazepine (remimazolam) and ketamine with unsecured airway
  3. Total intravenous anaesthesia with secured airway (arm TIVA): continuous propofol infusion using target controlled infusion (TCI) and short acting opioid boluses - sufentanil
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm P (Active Comparator): Patients in arm P will be administered 2-3 mg midazolam IV before the beginning of the procedure, 5-10 mcg sufentanil IV and a loading dose of propofol 0,8-1,0 mg/kg in 2-5 minutes before the start of the ablation phase. During the procedure, boluses of 0,5 mg/kg propofol will be repeated as needed, in case of inappropriate analgosedation, boluses of midazolam and/or sufentanil can also 0be repeated.
  Interventions: Drug: Propofol
- Arm R (Experimental): Patients in arm R will be administered 2,5 mg loading dose of remimazolam followed by continuous infusion at 0,5 mg/h/kg of ideal body weight (IBW, calculated using the Miller formula) and a dose of ketamine 1 mg/kg IBW 2-5 minutes before the beginning of the ablation phase. In case of inadequate sedation depth, a bolus of 2,5 mg remimazolam can be repeated as needed. If the patient shows signs of pain or discomfort, a single dose of ketamine - 0,5 mg/kg IBW - will be administered, followed by a bolus of 5-10 mcg sufentanil if needed. The continuous infusion will be terminated as the last ablation pulses are delivered.
  Interventions: Drug: Remimazolam
- Arm TIVA (Total Intravenous Anesthesia) (Active Comparator): Patients randomised in arm TIVA will be administered light analgosedation with spontaneous ventilation for the first part of the procedure. The analgosedation will be induced and maintained with bolus of 5 mcg sufentanil IV and propofol infusion dosed by TCI system (the target plasma concentration for propofol 1-2 mcg/ml). Before the beginning of the ablation phase, general anesthesia will be induced with one bolus of 5-10 mcg sufentanil (the TCI target 3-7 mcg/ml for induction and 3-5 mcg/ml for the rest of the procedure), and a bolus of rocuronium 0,2-0,4 mg/kg IBW. Then, the airways will be secured with a laryngeal mask (LMA), the patient ventilated (0,4 - 0,45 FiO2, the target EtCO2 30 - 45 mmHg). After the last ablation pulse is delivered, infusion of propofol will be ceased and LMA extracted at the return of consciousness, muscle strength and sufficient spontaneous ventilation. If residual muscle relaxation occurs, sugammadex will be administered.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — analgosedation without secured airway
  Arms: Arm R
Drug: Propofol — analgosedation with secured airway
  Arms: Arm P
Drug: Propofol — TIVA with secured airway
  Arms: Arm TIVA (Total Intravenous Anesthesia)

SUMMARY:
A prospective single blinded (subject blinded) 1:1:1 randomised control trial with three parallel arms testing superiority of analgosedation regimen based on remimazolam and total intravenous anesthesia over propofol based analgosedation. The primary composite endpoint consists of hypoxaemia, hypotension, or hypertension requiring intervention.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation (AF) (paroxysmal, persistent or long standing persistent) with indication for catheter ablation
* Age above 18 years
* Capacity to give informed consent

Exclusion Criteria:

* Heart failure (NYHA III-IV), irrespective of left ventricular ejection fraction
* Left ventricular ejection fraction < 20%
* Significant valvulopathy (moderate or severe aortic stenosis, severe mitral regurgitation, severe aortic regurgitation, moderate and severe mitral stenosis, severe tricuspid regurgitation)
* Obstructive sleep apnoea syndrome (AHI >30)
* Low oxygen saturation (<93%) at baseline
* High aspiration risk (hiatal hernia, gastroesophageal reflux disease on chronic pharmacotherapy)
* Hypersensitivity to the study drugs
* Chronic kidney disease (stage 4 and 5 of CKD), liver cirrhosis
* Anticipated difficult airways
* ASA (American Society of Anaesthesiologists) score > 4
* Schizophrenia
* Epilepsy
* Other individual contraindications (will be reported in detail)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Primary composite endpoint (rate of hypoxaemia, hypotension, or hypertension events) | Procedure duration
  Composite endpoint consisting of the rate of (1) hypoxaemia events requiring intervention, (2) hypotension events requiring intervention or leading to the procedure interruption, or (3) hypertension events requiring intervention

SECONDARY OUTCOMES:
Total number of haemodynamic instability events (hypoxemia, hypotension, hypertension; defined above), each five minutes of a continuous instability counts as a new event, as well as an instability persisting despite an intervention | Procedure duration
Total number of: a) hypoxemia events hypoxaemia <85% (more than 60s) b) hypotension events = systolic blood pressure (SBP) < 85 mmHg (more than 60s) c) hypertension event = SBP > 200 mmHg (more than 60s) | Procedure duration
Total number of interventions a) jaw thrust b) nasopharyngeal airway administration c) LMA / orotracheal intubation d) increasing FiO2 (oxygen flow) e) hypotensive drugs administration f) vasoactive drugs administration (ephedrine, noradrenaline) | Procedure duration
Total procedural time | Procedure duration
Analgosedation depth by bispectral (BIS) monitoring: area under the curve of BIS index (measured every 3 minutes during the procedure) | Procedure duration
Procedural sedation quality | 12-24 hours after the procedure
  PROcedural Sedation Assessment Survey - a previously validated form
Difficult sedation score | Procedure duration
  1-10 scale (10 = the worst), reported by an anaesthesiologist
Operator's satisfaction score | Procedure duration
  1-10 scale (10 = the worst), reported by the operating physician
Total number of serious adverse events | From randomization until discharge
  death, cardiopulmonary resuscitation (chest compression or adrenaline administration), an emergency intubation or prolonged stay in intensive care unit
carbon dioxide partial pressure after the procedure | blood sample taken after the procedure (up to 10 minutes)
  partial pressure (kPa) of CO2 measured in an arterial blood sample
28-day serious adverese events | discharge to the day 28
  death, a condition related to the procedure requiring inpatient hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Kralovske Vinohrady, Prague, Czechia, Czechia

REFERENCES:
- [Derived] Sochorova V, Kunstatova V, Osmancik P, Duska F, Herman D, Waldauf P, Poviser L, Karch J, Znojilova L, Filipcova V, Hozmanova J, Vesela J, Hozman M. COOPERATIVE-PFA: A Three-Arm Randomized Controlled Trial. Circulation. 2025 Jul 22;152(3):150-159. doi: 10.1161/CIRCULATIONAHA.125.074427. Epub 2025 Apr 27. PMID 40287932